CLINICAL TRIAL: NCT02585479
Title: Systemic Chemotherapy VersusTranscatheter Arterial Chemoembolization As Palliative Chemotherapy in Patients With Advanced Hepatocellular Carcinoma(HCC)
Brief Title: Systemic Chemotherapy Versus Transcatheter Arterial Chemoembolization(TACE) for Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: It doesn't meet the requirements of randomized trials
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Liao, Director, Principal Investigator, Clinical Professor, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-C/Ahcc
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pirarubicin; Oxaliplatin; Ethiodized Oil; Gelatin Sponge, Absorbable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- systemic chemotherapy (Experimental): Pirarubicin 30mg/m2 intravenously on Day 1 and Oxaliplatin 100 mg/m2 intravenously on Day 2 every 3 weeks until disease progression or limiting toxicity.
  Interventions: Drug: Pirarubicin; Drug: Oxaliplatin
- Transcatheter Arterial Chemoembolization (Active Comparator): Lipiodol 5-10ml,Pirarubicin17mg/m2 and Oxaliplatin 30mg/m2 are infused through the right and left hepatic arteries,followed by embolization using Gelfoam every 4 weeks until disease progression or limiting toxicity.
  Interventions: Drug: Pirarubicin; Drug: Oxaliplatin; Drug: Lipiodol; Device: Gelfoam

INTERVENTIONS:
Drug: Pirarubicin — 1. Pirarubicin 30mg/m2 intravenously
  2. Pirarubicin17mg/m2 are infused through the right and left hepatic arteries
Drug: Oxaliplatin — 1. Oxaliplatin 100 mg/m2 intravenously
  2. Oxaliplatin 30mg/m2 are infused through the right and left hepatic arteries
  Other Names: Eloxatin
Drug: Lipiodol — Lipiodol 5-10ml infused through the right and left hepatic arteries
  Arms: Transcatheter Arterial Chemoembolization
Device: Gelfoam — Hepatic artery embolization with Gelfoam.
  Arms: Transcatheter Arterial Chemoembolization

SUMMARY:
The purpose of this study is to determine that systemic chemotherapy is superior to transcatheter arterial chemoembolization in prolonging progression-free survival（PFS） in patients with Advanced Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were age 18 to 75 years;
* The patients had histologically, cytologically,or clinically diagnosed unresectable HCC;and were ineligible for local invasive treatment. Clinically diagnosed patients had to have: (1) evidence of HBV or HCV with hepatic cirrhosis; (2) a-fetoprotein levels 400g/L; and (3) morphologic evidence of hypervascular liver tumor. Patients had to have at least one measurable lesion according to RECIST (version 1.0; ≥2 cm on computed tomography [CT]; 1 cm on spiral CT or magnetic resonance imaging). Lesions that had undergone previous interventional or local therapy were not considered measurable lesions.
* ECOG score≤2;
* life expectancy 3 months;
* Barcelona Clinic liver cancer (BCLC) stage B or C disease;
* Child-Pugh stage A or B disease;
* Adequate organ and marrow function, with neutrophil count≥1.5X10e9/L, platelet count≥75×10e9/L, AST or ALT﹤2.5×upper limit of normal (ULN), total bilirubin <1.5×ULN, international normalized ratio <1.5;normal baseline left ventricular ejection fraction_lower limit of normal for the institution. Patients with AST and ALT<5 ×ULN could be recruited if total bilirubin was in the normal range.
* Patients had to provide signed informed consent to participate.

Exclusion Criteria:

* documented allergy to lipoidal or other study drugs; any previous treatment before random assignment;
* Previous liver transplantation;
* concomitant use of any other anticancer therapy, including interferon alfa and herbal medicine approved by the local authority to be used as anticancer medicine (except palliative radiotherapy to a nontarget lesion);
* CNS metastasis;
* Other serious illness or medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free-Survival | 3 months

SECONDARY OUTCOMES:
Objective response rate | 3 months
Overall survival | 6 months and 12 months
Time-to-Progression | 3 months
Time-to-Progression within liver | 3 months
Time-to-Progression outside the liver | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lequn Li, PhD, Study Director — Affiliated Tumor Hospital, Guangxi Medical University

REFERENCES:
- [Background] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077
- [Background] Li L, Sun F, Chen AJ, Li XY, Hu MD, Ran JH, Tang JH. [Capecitabine combined with TACE for advanced liver cancer]. Zhonghua Zhong Liu Za Zhi. 2004 Sep;26(9):565-6. Chinese. PMID 15555291
- [Background] Mabed M, Esmaeel M, El-Khodary T, Awad M, Amer T. A randomized controlled trial of transcatheter arterial chemoembolization with lipiodol, doxorubicin and cisplatin versus intravenous doxorubicin for patients with unresectable hepatocellular carcinoma. Eur J Cancer Care (Engl). 2009 Sep;18(5):492-9. doi: 10.1111/j.1365-2354.2008.00984.x. PMID 19453695